CLINICAL TRIAL: NCT01126450
Title: A Phase I, Open-Label Study To Determine The Maximum Tolerated Dose (Mtd) Of The Combination Of Lenalidomide And Cetuximab, And To Evaluate The Efficacy Of This Combination In Subjects With Wild Type K-Ras Metastatic Colorectal Carcinoma
Brief Title: Lenalidomide and Cetuximab in Treating Patients With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual,loss of funding and results from EU study showing drug ineffective.
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE8208; NCI-2010-01202 (Other: National Cancer Institute); CASE8208 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2010-05-18; First posted 2010-05-19 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Lenalidomide; Cetuximab; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral lenalidomide once daily on days 1-28 and cetuximab IV once weekly over 1-2 hours on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lenalidomide; Biological: cetuximab; Other: mutation analysis; Other: polymerase chain reaction; Genetic: polymorphism analysis

INTERVENTIONS:
Drug: lenalidomide — Given orally
  Other Names: CC-5013; IMiD-1; Revlimid
Biological: cetuximab — Given IV
  Other Names: Anti-EGFR Monoclonal Antibody; C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
Other: mutation analysis — Correlative studies
Other: polymerase chain reaction — Correlative studies
  Other Names: PCR
Genetic: polymorphism analysis — Correlative studies

SUMMARY:
RATIONALE: Lenalidomide may stop the growth of tumor cells by blocking blood flow to the tumor. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving lenalidomide together with cetuximab may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of lenalidomide when given together with cetuximab in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD).

SECONDARY OBJECTIVES:

I. To further explore the safety and efficacy profile.

OUTLINE:

This is a dose-escalation study of lenalidomide.

Patients receive oral lenalidomide once daily on days 1-28 and cetuximab IV once weekly over 1-2 hours on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion

* Wild type metastatic colorectal cancer that failed (progressed, refused or not tolerated) on at least two treatment regimens including a fluoropyrimidine, oxaliplatin and irinotecan with or without bevacizumab
* At least 28 days must have lapsed since completion of prior chemotherapy
* Subjects must understand and voluntarily sign an informed consent document
* Subjects must be able to adhere to the study visit schedule and other protocol requirements
* Histological or cytological diagnosis of colorectal carcinoma
* Radiographic or clinical evidence of a measurable disease (by RECIST criteria)
* Subjects must have received prior treatment with at least 2 prior regimens of therapy
* ECOG performance status of =< 1
* Anticipated survival >= 3 months
* Must agree to also take low dose aspirin (or other anticoagulation if unable to take ASA) while receiving study drug and for 30 days after study drug is discontinued
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test within 10-14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide; FCBP must also agree to ongoing pregnancy testing
* Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy

Exclusion

* Pregnant or lactating females
* CrCl < 50 mL/min by Cock-Croft and Gault
* Any serious medical condition or psychiatric illness that places the subject at an unacceptable risk for study participation or would prevent the subject from signing the informed consent
* Use of any cytotoxic chemotherapy within 28 days of study Day 1
* Use of therapeutic radiation =< 14 days prior to study Day 1
* Use of thalidomide, or structurally related compounds or biologic response modifier therapy within 14 days of study Day 1
* Prior desquamating rash while taking thalidomide, or structurally related compound therapy
* Prior >= Grade 2 allergic reaction to thalidomide or structurally related compounds
* Any prior use of Lenalidomide
* Subjects may have received prior thalidomide
* Known or suspected brain metastases
* Concurrent use or anticipated use of any other anti-cancer agents (except for stable dose steroid use for control of metastases symptoms) during participation in this study
* Absolute Neutrophil Count =< 1500/mm^3 (or 1.5 X10^9/L)
* Platelet Count =< 100,000/mm^3 (or 100 X 10^9/L)
* Hemoglobin < 8.0 g/dL
* Total Bilirubin > 2.0mg/dL
* Alanine Aminotransferase (ALT/SGPT) >= 3 x upper limit of normal (ULN)
* Aspartate Aminotransferase (AST/SGOT) >= 3 x upper limit of normal (ULN)
* Peripheral neuropathy >= Grade 2
* Active infection
* Subjects with an infection that is amenable to curative treatment may be eligible for screening once the infection has been treated, cured and not recurred for at least 14 days
* Uncontrolled hyper- or hypo- calcemia, glycosemia or thyroidism
* Arterial or venous thrombotic event in the preceding six months
* Known history of HIV infection
* Active viral hepatitis who is on active treatment
* No other malignancies, other than previously treated non-melanoma skin cancer or carcinoma insitu of the cervix or breast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-10; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety / Tolerability (type, frequency, severity, and relationship of adverse events to study drug) | Courses repeat every 28 days in the absence of unacceptable toxicity.

SECONDARY OUTCOMES:
Time to progression of disease | Courses repeat every 28 days in the absence of disease progression .
Tumor response according to RECIST | at the end of Cycle 2 and every 56 days thereafter until tumor progression
Lab correlatives (FCGRIIa and FCGRIIIa polymorphisms, K-Ras and B-Raf mutations) | Tissue collection less than or equal to 28 days prior to day 1 of therapy
  FCGR2a and FCGR3a polymorphisms, K-Ras and B-Raf mutations in patient specimens (paraffin embedded formaldehyde fixed tissues) will be identified.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kim, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States